CLINICAL TRIAL: NCT06461364
Title: Evaluation of Cuspal Deflection and Fracture Resistance of Different Bulk-fill Restorations and Their Clinical Performance in Class II Cavities
Brief Title: Clinical Performance of Bulk-fill Restorations in Class II Cavities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Egymedicalpedia (Industry)
Collaborators: Al-Azhar University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Walaa Hassan
Record Dates: First submitted 2024-06-09; First posted 2024-06-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Cavity, Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (Experimental): About 10 participants faced Self-adhesive composite (Surefil one)
  Interventions: Procedure: Assessment of cuspal deflection of bulk-fill restorations
- Group B (Experimental): About 10 participants faced Viscalor
  Interventions: Procedure: Assessment of cuspal deflection of bulk-fill restorations
- Group C (Experimental): About 10 participants faced Equiaforte
  Interventions: Procedure: Assessment of cuspal deflection of bulk-fill restorations

INTERVENTIONS:
Procedure: Assessment of cuspal deflection of bulk-fill restorations — To assess the performance of bulk-fill restorations on premolar teeth in class II cavities using some selected FDI criteria, a total sample size of 30 (10 for each group test) will be sufficient to detect: an effect size of 1.22 at a power (1-β error) of 0.8 and using a two-sided hypothesis test and a significance level (α error) 0.05 for data. Two teeth will be added to each group to compensate drop out samples.

SUMMARY:
Direct composite resin restorations are considered an essential treatment option in the dental clinic because of increasing the demands for esthetics. These materials are primarily used as anterior and posterior filling materials for the restoration of dental caries, crown fractures, tooth wear, and congenital defects.

DETAILED DESCRIPTION:
It has been reported that the polymerization shrinkage and its associated contraction stress are the greatest limitation in the use of resin-based composite (RBC) as a restorative material for posterior teeth.

Shrinkage stress that is generated due to the polymerization reaction is known as a multifaceted complicated condition. There are many factors aiding to development of the rate of shrinkage stress such as material formulation, degree of conversion, polymerization kinetics, flow capacity in the early stages of the curing reaction, and elastic modulus of the material itself.

Shrinkage stress appear in the form of several manifestations as cuspal movement which can result in enamel micro cracks, cervical marginal gaps, creating postoperative sensitivity, discoloration of the margins, recurrent caries, breakages of the restoration and finally replacement of composite restorations.

New types of restorative materials called bulk-fill restorative materials have been introduced to reduce time required for placement. These materials can be placed in bulk layer up to 4-5mm with adequate polymerization and low polymerization shrinkage stress. However, little information is available regarding the effect of these restorative materials on cuspal deflection.

The first thermoviscous bulk-fill composite, has the viscosity of a flowable composite and the sculptability of a packable composite all in a single material. Prior to placement, this material is warmed in a modified caps warmer. Bulk-fil composite satisfies the sealing of the proximal box as well as attains the desired anatomy in a single bulk-cure product in class II restorations.

Cuspal deflection is a common biomechanical phenomenon that occurs in teeth restored with composite resin-based materials and represents the interaction between polymerization stress of material and the compliance of remaining tooth structure, which may cause failure during composite curing or act as a preloading, facilitating tooth fracture under occlusal loads. Cuspal deflection can be perceived clinically by the patient as postoperative sensitivity.

The fracture of teeth is a common dental problem. Many factors such as tooth anatomy contribute to cusp fracture; however, cavity preparation procedures seem to be the major cause of most cuspal fractures. Posterior teeth, particularly premolars, have an anatomic shape that makes them more likely to fracture under occlusal load, whereas sound teeth are rarely fracture under normal masticatory function. Several studies have emphasized the importance of maintaining dental structure to preserve the strength of remaining tooth. Generally, the wider the involvement by caries or cavity preparation, the weaker the tooth.

The FDI criteria-based proposal allows to classify the evaluation of dental restorations, according to functional, biological and aesthetic categories. Their use was thus recommended in clinical trials assessing dental restorations in terms of materials, operative technique/intervention, as well as in clinical practice to determine whether a restoration should be maintained, repaired or replaced. One study compared the FDI criteria and the traditional United States Public Health Service (USPHS; also known as 'Ryge criteria') criteria for the evaluation of dental restorations.

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the study must be with at least two proximal caries teeth of ICDAS score 4.
* Patients with moderate and high caries risk index.
* Carious lesions will be standardized by means of clinical and radiographic examinations performed before the procedures.
* At least two permanent molars at one side requiring class ii caries lesions, with at least one neighboring tooth and in occlusion with antagonistic teeth.
* Moderate to large size cavities that extended into dentine, while maintain natural tooth contour.
* Absence of tooth mobility, tenderness, severe pain or pre-operative sensitivity.
* Normal occlusion relation with normal dentition

Exclusion Criteria:

* Teeth with deep dentinal lesions with pulpal involvement, abscess, pain or swelling
* Developmental disorders and adjacent soft tissue lesions.
* Patients with systemic illness will be excluded

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-07-20 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-25 (Actual)

PRIMARY OUTCOMES:
FDI criteria Esthetic | from 3 months to 12 months
  evaluated surface luster and surface staining
FDI criteria Functional | from 3 months to 12 months
  evaluated fracture of material and retention,occlusal contour and wear
FDI criteria Biological | from 3 months to 12 months
  Biological evaluated post operative hypersensitivity and recurrence caries

CONTACTS AND LOCATIONS:
Overall Officials: Wael Essam Jamil, Professor, Study Chair — Al-Azhar Faculty of Dentistary for girls
Locations (1):
- Faculty of Dentistary - Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No